CLINICAL TRIAL: NCT00121550
Title: The Effect of Clarithromycin on Mortality and Morbidity in Patients With Ischemic Heart Disease - a Randomized, Placebo Controlled, Double Blinded, Multicentre, Clinical Trial
Brief Title: The CLARICOR Trial: Effect of Clarithromycin on Mortality and Morbidity in Patients With Ischemic Heart Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Copenhagen Trial Unit, Center for Clinical Intervention Research (Other)
Collaborators: Danish Heart Foundation (Other); Copenhagen Hospital Corporation (Other); The Danish Medical Research Council (Other); The 1991 Pharmacy Foundation (Other); Abbott (Industry)
Responsible Party: Principal Investigator, Christian Gluud, MD, DMSc, Copenhagen Trial Unit, Center for Clinical Intervention Research
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1997-08-DP-42-RKF-13 CLARICOR;; REC: KF01-076/99; DDPA: 2001-41-1496,; DMA: 2612-975
Record Dates: First submitted 2005-07-13; First posted 2005-07-21 (Estimated); Last update posted 2016-08-11 (Estimated); Status verified 2016-08

CONDITIONS: Heart Disease; Cardiovascular Disease
Keywords: Coronary heart disease; Clarithromycin; Macrolides; Cardiovascular mortality; Chlamydia pneumoniae
MeSH Terms: conditions — Heart Diseases; Cardiovascular Diseases; Coronary Disease | interventions — Clarithromycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Clarithromycin (Experimental): Clarithromycin is a lipophilic semi-synthetic macrolide antibiotic. The lipophilic nature of the drug allows it to easily penetrate into body fluids and tissues and accumulate intracellularly. Side effects are few, apart from trivial gastrointestinal complaints, and severe side effects are rarely observed during standard treatment.
  Interventions: Drug: clarithromycin
- Placebo (Placebo Comparator): Placebo comparator
  Interventions: Drug: clarithromycin

INTERVENTIONS:
Drug: clarithromycin

SUMMARY:
A growing body of evidence links Chlamydia pneumoniae to the progression of coronary heart disease. The purpose of this study is to determine the positive and negative effect of 14 days treatment with clarithromycin 500 mg daily in patients already suffering from stable coronary heart disease. The participants will be followed for at least two years after the treatment.

Abbott Laboratories supplied Clarithromycin and placebo tablets.

DETAILED DESCRIPTION:
Basic science suggests a fundamental role for inflammation in mediating all stages of coronary heart disease (CHD), and a large number of clinical studies have reported an association between markers of inflammation and CHD. Consequently, infectious agents have been proposed as promoters of atherosclerosis and/or acute coronary syndrome (ACS). Many studies have suggested a relation between Chlamydia pneumoniae (C. pneumoniae) infection and CHD, and C. pneumoniae has been demonstrated in atherosclerotic tissue.

Macrolide antibiotics are effective in eradication of C. pneumoniae from atherosclerotic plaques. Two small trials showed significant beneficial effects of macrolides on cardiovascular morbidity in patients with ACS. To corroborate and extend these findings, we undertook a randomised, placebo-controlled trial with clarithromycin in patients with stable CHD in order to test the hypothesis that intervention with a macrolide would reduce cardiovascular risk with regard to mortality and morbidity.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 18 to 85 years and
* previous acute myocardial infarction (AMI) or
* previous or present angina pectoris and
* signed informed concent

Exclusion Criteria:

* AMI or unstable angina pectoris within the last three months
* revascularisation (PTCA or CABG) within the preceding six months
* severe heart failure (New York Heart Association (NYHA) functional class IV)
* known impaired renal or hepatic function
* active malignancy
* intolerance to macrolides
* treatment with methylxanthines, carbamazepine, cisapride, astemizole, terfenadine, or coumarin anticoagulants
* earlier inclusion in the CLARICOR Trial or participation in another drug trial within four weeks
* participation in other clinical trials within one month before this trial
* individuals incapable of managing own affairs or not able to sign written consent
* lack of written consent
* women of childbearing age not using reliable contraceptives
* breast feeding women

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4372 (Actual)
Dates: Start 1999-10; Primary Completion 2000-04 (Actual); Study Completion 2002-09 (Actual)

PRIMARY OUTCOMES:
Composite consisting of: death regardless of cause
non-fatal AMI or
unstable angina pectoris whichever occurred first

SECONDARY OUTCOMES:
Composite of: cardiovascular death
non-fatal AMI or
unstable angina pectoris whichever occurred first

CONTACTS AND LOCATIONS:
Overall Officials: Christian Jespersen, DMSc, Study Chair — Department of Cardiology Y, Bispebjerg Hospital, Bispebjerg Bakke 23, DK 2400 Copenhagen NV, Denmark.; Christian Gluud, DMSc, Principal Investigator — Copenhagen Trial Unit, Center of Clinical Intervention Research, Rigshospitalet, Copenhagen University Hospital, Blegdamsvej 9, DK-2100 Copenhagen
Locations (6):
- Denmark (6):
  - Copenhagen Trial Unit, Center for Clinical Intervention Research, Rigshospitalet, Copenhagen University Hospital, Blegdamsvej 9, Copenhagen
  - H:S Rigshospitalet, Copenhagen
  - H:S Amager Hospital, Copenhagen
  - H:S Bispebjerg Hospital, Copenhagen
  - H:S Frederiksberg Hospital, Frederiksberg
  - H:S Hvidovre Hospital, Hvidovre

REFERENCES:
- [Background] Hansen S, Als-Nielsen B, Damgaard M, Helø OH, Petersen L, Jespersen CM. Intervention with clarithromycin in patients with stable coronary heart disease. The CLARICOR Trial Design. Heart Drug 2001;1:14-9.
- [Result] Jespersen CM, Als-Nielsen B, Damgaard M, Hansen JF, Hansen S, Helo OH, Hildebrandt P, Hilden J, Jensen GB, Kastrup J, Kolmos HJ, Kjoller E, Lind I, Nielsen H, Petersen L, Gluud C; CLARICOR Trial Group. Randomised placebo controlled multicentre trial to assess short term clarithromycin for patients with stable coronary heart disease: CLARICOR trial. BMJ. 2006 Jan 7;332(7532):22-7. doi: 10.1136/bmj.38666.653600.55. Epub 2005 Dec 8. PMID 16339220
- [Derived] Winkel P, Hilden J, Jakobsen JC, Lindschou J, Jensen GB, Kjoller E, Sajadieh A, Kastrup J, Kolmos HJ, Larsson A, Arnlov J, Bjerre M, Gluud C. A screening method to spot biomarkers that may warn of serious events in a chronic disease - illustrated by cardiological CLARICOR trial data. Clin Chem Lab Med. 2021 Aug 12;59(11):1852-1860. doi: 10.1515/cclm-2021-0333. Print 2021 Oct 26. PMID 34384145
- [Derived] Winkel P, Jakobsen JC, Hilden J, Jensen GB, Kjoller E, Sajadieh A, Kastrup J, Kolmos HJ, Iversen KK, Bjerre M, Larsson A, Arnlov J, Gluud C. Prognostic value of 12 novel cardiological biomarkers in stable coronary artery disease. A 10-year follow-up of the placebo group of the Copenhagen CLARICOR trial. BMJ Open. 2020 Aug 20;10(8):e033720. doi: 10.1136/bmjopen-2019-033720. PMID 32819979
- [Derived] Bjerre M, Hilden J, Winkel P, Jensen GB, Kjoller E, Sajadieh A, Kastrup J, Kolmos HJ, Larsson A, Arnlov J, Jakobsen JC, Gluud C. Serum osteoprotegerin as a long-term predictor for patients with stable coronary artery disease and its association with diabetes and statin treatment: A CLARICOR trial 10-year follow-up substudy. Atherosclerosis. 2020 May;301:8-14. doi: 10.1016/j.atherosclerosis.2020.03.030. Epub 2020 Apr 4. PMID 32289619
- [Derived] Schroder J, Jakobsen JC, Winkel P, Hilden J, Jensen GB, Sajadieh A, Larsson A, Arnlov J, Harutyunyan M, Johansen JS, Kjoller E, Gluud C, Kastrup J. Prognosis and Reclassification by YKL-40 in Stable Coronary Artery Disease. J Am Heart Assoc. 2020 Mar 3;9(5):e014634. doi: 10.1161/JAHA.119.014634. Epub 2020 Mar 2. PMID 32114892
- [Derived] Winkel P, Jakobsen JC, Hilden J, Lange T, Jensen GB, Kjoller E, Sajadieh A, Kastrup J, Kolmos HJ, Larsson A, Arnlov J, Gluud C. Predictors for major cardiovascular outcomes in stable ischaemic heart disease (PREMAC): statistical analysis plan for data originating from the CLARICOR (clarithromycin for patients with stable coronary heart disease) trial. Diagn Progn Res. 2017 Mar 29;1:10. doi: 10.1186/s41512-017-0009-y. eCollection 2017. PMID 31093541
- [Derived] Winkel P, Jakobsen JC, Hilden J, Jensen G, Kjoller E, Sajadieh A, Kastrup J, Kolmos HJ, Larsson A, Arnlov J, Gluud C. Prognostic value of routinely available data in patients with stable coronary heart disease. A 10-year follow-up of patients sampled at random times during their disease course. Open Heart. 2018 Sep 5;5(2):e000808. doi: 10.1136/openhrt-2018-000808. eCollection 2018. PMID 30228904
- [Derived] Carlsson AC, Ruge T, Kjoller E, Hilden J, Kolmos HJ, Sajadieh A, Kastrup J, Jensen GB, Larsson A, Nowak C, Jakobsen JC, Winkel P, Gluud C, Arnlov J. 10-Year Associations Between Tumor Necrosis Factor Receptors 1 and 2 and Cardiovascular Events in Patients With Stable Coronary Heart Disease: A CLARICOR (Effect of Clarithromycin on Mortality and Morbidity in Patients With Ischemic Heart Disease) Trial Substudy. J Am Heart Assoc. 2018 Apr 23;7(9):e008299. doi: 10.1161/JAHA.117.008299. PMID 29686027
- [Derived] Kjoller E, Hilden J, Winkel P, Galatius S, Frandsen NJ, Jensen GB, Fischer Hansen J, Kastrup J, Jespersen CM, Hildebrandt P, Kolmos HJ, Gluud C; CLARICOR Trial Group. Agreement between public register and adjudication committee outcome in a cardiovascular randomized clinical trial. Am Heart J. 2014 Aug;168(2):197-204.e1-4. doi: 10.1016/j.ahj.2013.12.032. Epub 2014 May 4. PMID 25066559
- [Derived] Lyngbaek S, Winkel P, Gotze JP, Kastrup J, Gluud C, Kolmos HJ, Kjoller E, Jensen GB, Hansen JF, Hildebrandt P, Hilden J; CLARICOR Trial Group. Risk stratification in stable coronary artery disease is possible at cardiac troponin levels below conventional detection and is improved by use of N-terminal pro-B-type natriuretic peptide. Eur J Prev Cardiol. 2014 Oct;21(10):1275-84. doi: 10.1177/2047487313492099. Epub 2013 May 30. PMID 23723326
- [Derived] Winkel P, Hilden J, Fischer Hansen J, Hildebrandt P, Kastrup J, Kolmos HJ, Kjoller E, Jespersen CM, Gluud C, Jensen GB; CLARICOR Trial Group. Excess sudden cardiac deaths after short-term clarithromycin administration in the CLARICOR trial: why is this so, and why are statins protective? Cardiology. 2011;118(1):63-7. doi: 10.1159/000324533. Epub 2011 Mar 26. PMID 21447948
- [Derived] Harutyunyan MJ, Mathiasen AB, Winkel P, Gotze JP, Hansen JF, Hildebrandt P, Jensen GB, Hilden J, Jespersen CM, Kjoller E, Kolmos HJ, Gluud C, Kastrup J; CLARICOR Trial Group. High-sensitivity C-reactive protein and N-terminal pro-B-type natriuretic peptide in patients with stable coronary artery disease: a prognostic study within the CLARICOR trial. Scand J Clin Lab Invest. 2011 Feb;71(1):52-62. doi: 10.3109/00365513.2010.538081. Epub 2010 Nov 25. PMID 21108561
- [Derived] Jensen GB, Hilden J, Als-Nielsen B, Damgaard M, Hansen JF, Hansen S, Helo OH, Hildebrandt P, Kastrup J, Kolmos HJ, Kjoller E, Lind I, Nielsen H, Petersen L, Jespersen CM, Gluud C; CLARICOR Trial Group. Statin treatment prevents increased cardiovascular and all-cause mortality associated with clarithromycin in patients with stable coronary heart disease. J Cardiovasc Pharmacol. 2010 Feb;55(2):123-8. doi: 10.1097/FJC.0b013e3181c87e37. PMID 19920766
- [Derived] Jespersen CM, Kolmos HJ, Frydendall N, Hilden J, Gluud C, Hansen JF; CLARICOR Trial Group. Compliance with and short-term adverse events from clarithromycin versus placebo in patients with stable coronary heart disease: the CLARICOR trial. J Antimicrob Chemother. 2009 Aug;64(2):411-5. doi: 10.1093/jac/dkp190. Epub 2009 May 28. PMID 19477891